CLINICAL TRIAL: NCT06678503
Title: ADDING CORE STABILITY EXERCISES TO CONVENTIONAL PROGRAM IN ATHLETES WITH CHRONIC ANKLE INSTABILITY
Brief Title: Core Stability Traning Exercises in Chronic Ankle Instability in Atheletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, abanoub malak latif, Physical therapist, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005346
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Chronic Ankle Instability and Balance
Keywords: Core stability Balance CAI Atheletes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple ( Participant, Care provider, outcomes Assessor )
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): 1. Single legged stance:
  2. Single-legged stance on the balance board
  3. Single legged hop
  4. Quadrant Hop:
  5. Single legged Ball Catch:
  6. Hop ups and downs:
  Interventions: Other: balance exercise
- Experimental Group (Experimental): Participants Will perform the same exercises in addition to core exercises
  The core exercises will include 12 different exercises:
  Week 1 :
  1. Abdominal Drawing In
  2. Abdominal Drawing in with alternating lower limb movement
  3. Pelvic tilting with standing
  4. Forward lunge
  Week 2 :
  1. Bracing with bridging
  2. Curl up with bracing
  3. Quadruped with bracing
  4. Side plank with knee flexed
  Week 3 :
  1. Bracing with straight leg raising
  2. Quadruped leg lift with bracing
  3. Bridging with bracing on a Swiss ball
  4. Side plank with the knee extended
  Week 4 :
  1. Alternate arm and leg raise from quadruped
  2. Abdominal drawing in with a squat against a wall
  3. Single limb deadlift
  4. Squat with overhead sustained lift
  Interventions: Other: balance exercise; Other: Core stability exercises

INTERVENTIONS:
Other: balance exercise — Balance exercises are physical activities designed to improve stability, coordination, and posture by challenging the body's ability to maintain an upright position. These exercises target the muscles and systems involved in balance, particularly the core, legs, and the sensory systems (like vision and proprioception).
Other: Core stability exercises — Core stability exercises are physical activities designed to improve the strength, endurance, and coordination of the muscles that support and stabilize the spine, pelvis, and torso. These exercises specifically target the muscles of the abdomen, lower back, hips, and pelvis, collectively referred to as the "core." The goal is to enhance overall posture, prevent injury, and improve performance in daily activities or sports by increasing the body's ability to stabilize itself during movement.
  Arms: Experimental Group

SUMMARY:
To study the effect of adding Core stability exercise to the conventional Program of Chronic ankle instability on balance, Functional instability, and Performance in athletes with CAI

DETAILED DESCRIPTION:
Chronic Ankle Instability (CAI) is a prevalent and debilitating condition that afflicts a considerable portion of the population (Al Adal et al.,2020) it is a condition characterized by repetitive episodes or perceptions of the ankle giving way; ongoing symptoms such as pain, weakness, or reduced ankle range of motion (ROM); diminished self-reported function; and recurrent ankle sprains that persist for more than 1 year after the initial injury (Gribble et al.,2013).

Purpose of the Study To study the effect of adding Core stability exercise to the conventional Program of Chronic ankle instability on balance, Functional instability, and Performance in athletes with CAI Methods:Triple Blinded RCT (Blinded: Participants, Research Assistant (for assessment of patient pre- and post-intervention) and statistician) Results :An unpaired t-test will be conducted for comparison of age, weight, and height between groups.

* Chi-squared test will be conducted for comparison of sex distribution between groups
* Mixed MANOVA will be conducted to compare the effect of time (pre versus post) and the effect of treatment (between groups), as well as the interaction between time and treatment on dependent variables.
* The level of significance for all statistical tests will be set at p < 0.05.
* All statistical measures will be performed through the statistical package for social sciences (SPSS) version 25 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Athletes having a history of chronic lateral ankle sprain during the offseason period.

  2. Patients aged between 19-30 years, with BMI ranging between (18.5-29.5kg/m2).

  3. Patients having unilateral CAI with the diagnosis to be based on the criteria described by the International Ankle Consortium for enrolling patients of CAI in controlled research (Gribble et al., 2014) as follows:
  1. A history of at least one significant ankle sprain (the initial sprain must have occurred at least more than 3 months prior to study enrollment, at least one interrupted day of desired physical activity.
  2. Participants should report at least 2 episodes of giving way and/or recurrent sprain and/or feelings of instability in the 6 months prior to study enrollment.
  3. Self-reported ankle instability should be confirmed using a validated ankle instability questionnaire, CAIT>24.

     Exclusion Criteria:
* Those with a history of spine, pelvis, and lower extremity injury, fracture, or surgery.

  2- Those with LBP that required medical or surgical intervention. 3- Those who participated in supervised or unsupervised ankle rehabilitation within 3 months before enrollment in the study.

  4- Having a history of an acute lower extremity injury in the 3 months before the study.

  5. Participation in formal rehabilitation in the 3 months before the study. 6. Having a history of lower extremity surgery or fracture that required alignment in the involved limb.

  7. Being diagnosed with neurologic dysfunction, such as multiple sclerosis, Parkinson's disease, or head injury.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Star Excursion Balance test | 4 weeks
  is a reliable functional test to evaluate dynamic postural control of the lower limb and distinguish CAI from copers and healthy individuals

SECONDARY OUTCOMES:
Functional Instability | 4 weeks
  The Cumberland Ankle Instability Tool assesses ankle instability during activities of daily living and sports and is valid and reliable for determining the presence of CAI
Functional Performance | 4 weeks
  Functional performance tests are dynamic measures used to assess general lower body function. These tests are helpful because they combine multiple components, such as muscular strength, neuromuscular coordination, and joint stability, which could be affected after joint injury.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy Yousef, Professor, Study Chair — Cairo University; Tarek Saad, Associate Professor, Study Director — Cairo University; Aya Ahmed Nada, PHD, Study Director — Pharos University in Alexandria

REFERENCES:
- [Background] Huang PY, Chen WL, Lin CF, Lee HJ. Lower extremity biomechanics in athletes with ankle instability after a 6-week integrated training program. J Athl Train. 2014 Mar-Apr;49(2):163-72. doi: 10.4085/1062-6050-49.2.10. Epub 2014 Feb 25. PMID 24568224
- [Result] Herzog MM, Kerr ZY, Marshall SW, Wikstrom EA. Epidemiology of Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):603-610. doi: 10.4085/1062-6050-447-17. Epub 2019 May 28. PMID 31135209
- [Result] Hale SA, Fergus A, Axmacher R, Kiser K. Bilateral improvements in lower extremity function after unilateral balance training in individuals with chronic ankle instability. J Athl Train. 2014 Mar-Apr;49(2):181-91. doi: 10.4085/1062-6050-49.2.06. Epub 2014 Feb 25. PMID 24568231
- [Result] Hall EA, Chomistek AK, Kingma JJ, Docherty CL. Balance- and Strength-Training Protocols to Improve Chronic Ankle Instability Deficits, Part I: Assessing Clinical Outcome Measures. J Athl Train. 2018 Jun;53(6):568-577. doi: 10.4085/1062-6050-385-16. Epub 2018 Jul 5. PMID 29975573
- [Result] Hiller CE, Nightingale EJ, Raymond J, Kilbreath SL, Burns J, Black DA, Refshauge KM. Prevalence and impact of chronic musculoskeletal ankle disorders in the community. Arch Phys Med Rehabil. 2012 Oct;93(10):1801-7. doi: 10.1016/j.apmr.2012.04.023. Epub 2012 May 7. PMID 22575395